CLINICAL TRIAL: NCT03490136
Title: Secular TRends in DiabEtes in India
Brief Title: Secular Trends in the Prevalence of Diabetes in India
Acronym: STRiDE-I
Status: Completed | Type: Observational
Sponsor: India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: IDRF-ARH-004
Record Dates: First submitted 2018-03-07; First posted 2018-04-06 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Type2 Diabetes; PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Series of epidemiological studies have been carried out by the research team since 1988 studying the changes in the prevalence of type 2 diabetes, prediabetes and associated risk factors. These studies have shown that the determinants to rising prevalence of diabetes vary among populations and with time. Comparative studies from the same region can help to understand the secular changes occurring in a specific population. In this proposal we intend to conduct a cross-sectional survey with varied levels of urbanisation and compare the findings with our earlier reported data to assess the degree of changes in dysglycaemic prevalences. The primary aim of the proposal is to study the secular changes and the prevalence of diabetes, prediabetes and associated cardio-metabolic risk factors with varying levels of urbanization.

A multi-stage random selection method will be used. Field workers will conduct an enumeration of the individuals above 20 years of age. In each location, streets will be randomly selected to have an equal representativeness from different socio-economic strata. All eligible family members of the selected households are invited for the survey. The study outcomes will be of relevance in public health research in modeling effective national healthcare policies.

ELIGIBILITY:
Inclusion Criteria:

Willing to participate and provide informed consent form.

Exclusion Criteria:

Age less than 20 years,cognitive impairment, unwilling to participate

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Households of selected families of a city, town and peri-urban village
Sampling Method: Non-Probability Sample
Enrollment: 9848 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of type 2 diabetes | Upto 18 months
  Prevalence of type 2 diabetes ,impaired fasting glucose and impaired glucose tolerance in a city, town and peri urban village in Southern India

SECONDARY OUTCOMES:
Secular trend in diabetes risk factors | Upto 18 months
Prevalence of cardiovascular risk factors | Upto 18 months
Prevalence of dysglycaemia in the young population aged ≤ 40 years | Upto 18 months
Prevalence of age-related hypertension in these regions | Upto 18 months
Changes in physical activity | Upto 18 months
Quality of diabetes care | Upto 18 months
Changes in dietary habits | Upto 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ambady Ramachandran, PhD DSc, Principal Investigator — President, India Diabetes Research Foundation
Locations (1):
- Dr.Ambady Ramachandran, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nanditha A, Susairaj P, Satheesh K, Raghavan A, Snehalatha C, Ramachandran A. The rising prevalence of type 2 diabetes among the youth in southern India-An ancillary analysis of the Secular TRends in DiabEtes in India (STRiDE-I) study. J Diabetes. 2024 Jul;16(7):e13576. doi: 10.1111/1753-0407.13576. PMID 38923743
- [Derived] Nanditha A, Snehalatha C, Satheesh K, Susairaj P, Simon M, Vijaya L, Raghavan A, Vinitha R, Ramachandran A. Secular TRends in DiabEtes in India (STRiDE-I): Change in Prevalence in 10 Years Among Urban and Rural Populations in Tamil Nadu. Diabetes Care. 2019 Mar;42(3):476-485. doi: 10.2337/dc18-1559. Epub 2019 Jan 18. PMID 30659076